CLINICAL TRIAL: NCT06699992
Title: Clinical Application and Usability of Blood Biomarkers As Screening Tool in Alzheimer Disease: a Validation Study
Acronym: BIOVALID-AD
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Istituto Superiore di Sanità (Other); Azienda Ospedaliera dei Colli (Other); Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other); A.O.U. Città della Salute e della Scienza (Other); Neurologia Arzignano AULSS8 Berica (Unknown); Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Marra Camillo, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6885
Record Dates: First submitted 2024-07-26; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-07

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Blood biomarkers quantification — Blood biomarkers quantification

SUMMARY:
Dementia caused by neurodegenerative diseases affects over 50 million people worldwide, Alzheimer's disease (AD) being the most common cause. As life expectancy increases, the prevalence of these diseases is expected to grow in coming decades, placing a significant social and economic burden on National Health Systems. AD is pathologically defined by two major hallmarks: amyloid-ß (Aß) accumulation in extracellular plaques, and hyperphosphorylated tau (p-tau) accumulation in intracellular neurofibrillary tangles. In recent decades, increased understanding of AD pathophysiology and technological advancements have allowed the development of new techniques providing an objective measure of AD pathological processes in vivo. Established biomarkers such as those obtained by cerebrospinal fluid (CSF) examination and positron emission tomography (PET) measures have been progressively introduced into clinical practice, consistently with the most recent NIA-AA diagnostic criteria. However, the widespread use of these methods remains limited due to their low availability, perceived invasiveness, high costs, and contraindications. Accordingly, there is a pressing need for costeffective biomarkers that can be less invasively obtained. Therefore, recent promising results in the development of ultrasensitive detection methods for blood biomarkers could facilitate a breakthrough in the field, simplifying and accelerating the diagnostic process of subjects with cognitive decline.

The main hypothesis of this study is that new plasma biomarkers of amyloidopathy, tauopathy, neurodegeneration, measured through a novel CLEIA methodology, may have the potential to change the diagnostic process of neurodegenerative diseases by reducing the need for unnecessary exams thus providing valuable information from a clinical and public health perspective. The larger availability and easier procedures for obtaining AD biomarkers from plasma, as compared to CSF, may also help to reduce territorial and economic disparities in reaching AD diagnosis. In addition, investigating biomarkers of neuroinflammation may provide new insights about the complex relations between AD pathogenetic processes, disease severity, and its prognosis.

This study aims to validate the reliability of biomarkers for AD and major neurodegenerative diseases, obtained from plasma instead of CSF. The findings will facilitate a paradigm shift in clinical practice toward the implementation of reliable and costeffective diagnostic tools that can be used not only for research purposes but also in clinical practice. This will also create new opportunities for population-based interventions, as well as future screening campaigns in primary care, reducing expenditures unnecessary investigations in individuals at low risk for dementia and delays in access to diagnosis and interventions that will slow cognitive decline in subjects at high risk for dementia. Thus, the validation of these novel biomarkers could have relevant positive economic and social implications for National Health Systems as well as for those personally affected by a neurodegenerative disease or their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* consecutive subjects with a clinical indication to undergo lumbar puncture for the determination of cerebrospinal fluid biomarkers of amyloidosis, tauopathy, and neurodegeneration during diagnostic assessments for cognitive impairment (as per clinical practice)
* informed consent form signed by patient or caregiver

Exclusion Criteria:

* Age under 50 or over 80 years
* Non-native Italian speakers
* History of previous or concurrent neurological diseases that could impact cognition (e.g., severe cerebrovascular accidents, brain tumors, traumatic injuries, etc.)
* History of major psychiatric disorders that could affect cognitive abilities
* History of alcohol use disorder
* Medical conditions that may interfere with cognitive functions (e.g., renal or hepatic failure, respiratory diseases, hypothyroidism, vitamin B12 deficiency, etc.)
* Uncompensated systemic disease with instability and significant organ failure
* Contraindications to lumbar puncture (e.g., presence of spinal malformations or current use of anticoagulant therapy)
* Previous or current participation in experimental studies involving amyloid-targeting agents

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will include subjects referred to the for an initial evaluation of cognitive disorders.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Accuracy of plasma biomarkers in identifying CSF biomarkers positive subjects | 2 years
  high agreement between CSF and plasma biomarkers values, equal to a value of AUC greater than 90%

SECONDARY OUTCOMES:
Plasma biomarkers cut offs | 2 years
  identification of accurate plasma biomarkers cut-offs (for single biomarkers of amyloidopathy, tauopathy, neurodegeneration and neuroinflammation and for combinations of the aforementioned markers) for distinguishing patients with AD from other forms of cognitive decline in a CCDD setting.
Validation of diagnostic performance | 2 years
  validation of the diagnostic performance of plasma biomarkers cut-offs previously established in a CCDD setting.
Prognostic performance | 2 years
  evaluation of the predictive value of blood biomarkers (for single biomarkers of amyloidopathy, tauopathy, neurodegeneration and neuroinflammation and for combinations of the aforementioned markers) for progression from MCI to AD in a community-based population.

CONTACTS AND LOCATIONS:
Overall Officials: Camillo Marra, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: No